CLINICAL TRIAL: NCT02897414
Title: Extended Release/Long Acting (ER/LA) Opioid Analgesics Risk Evaluation and Mitigation Strategy (REMS) Medical Examiner Surveillance Monitoring Protocol
Brief Title: ER/LA Opioid Analgesics - Surveillance Monitoring of State Medical Examiner Databases
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: ER/LA Opioid REMS Program Companies (RPC) (Industry)
Responsible Party: Sponsor
Other Study IDs: Assessment 5.5
Record Dates: First submitted 2016-08-10; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Opioid-related Disorders; Opioid Addiction; Narcotic Abuse; Drug Abuse
MeSH Terms: conditions — Opioid-Related Disorders; Narcotic-Related Disorders; Substance-Related Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective

GROUPS / COHORTS (5):
- Overall group of all ER/LA opioid excluding hydrocodone
  Interventions: Other: Surveillance of state medical examiner databases
- Each type of opioid that has an ER/LA opioid formulation
  Interventions: Other: Surveillance of state medical examiner databases
- Overall group that includes all prescription opioids except
  Interventions: Other: Surveillance of state medical examiner databases
- Comparator Group taking benzodiazepines
  Interventions: Other: Surveillance of state medical examiner databases
- Comparator Group taking IR hydrocodone
  Interventions: Other: Surveillance of state medical examiner databases

INTERVENTIONS:
Other: Surveillance of state medical examiner databases

SUMMARY:
In April 2011, the U.S. Food and Drug Administration (FDA) determined that a class-wide risk evaluation and mitigation strategy (REMS) for all extended-release (ER) and long-acting (LA) opioid medications was necessary to support national efforts to reduce serious adverse outcomes resulting from opioid abuse. This study will evaluate trends before and after the ER/LA REMS implementation for changes in mortality rates associated with prescription opioids utilizing state medical examiner databases from multiple states. Databases from 2005 through the most recent year available will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Fatalities associated with prescription opioids in several states during 2005-2015 (or later).

Exclusion Criteria:

* None

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Fatalities associated with prescription opioids as reported in State medical examiner databases from multiple states.
Sampling Method: Non-Probability Sample
Enrollment: 13015 (Estimated)
Dates: Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Rates of fatalities associated with prescription opioids per size of population covered by the surveillance systems | Review over period from January 2005 to 2016
Rates of fatalities associated with prescription opioids per number of prescriptions dispensed in the states | Review over period from January 2005 to 2016